CLINICAL TRIAL: NCT07166055
Title: The Effect of Therapeutic Dance on the Parameters of the International Classification of Functioning, Disability, and Health in Children With Functional Diversity
Brief Title: Effect of Dance on the Parameters of the ICF in Children With Functional Diversity
Acronym: DanceDiversity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, M Luz Sanchez, Professor, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-FIS-3495976
Record Dates: First submitted 2025-09-02; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Children With Disabilities
Keywords: dance therapy; motor impairment; dance movement therapy; neurological disease
MeSH Terms: conditions — Nervous System Diseases

STUDY DESIGN:
Intervention Model Description: Therapeutic dance
Who Masked: Outcomes Assessor
Masking Description: The researcher in charge of the statistical analysis is blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dance group (Experimental): Paticipants in this group will perform eight months of therapeutic dance classes (consisting of two one-hour sessions per week).
  Interventions: Other: Therapeutic dance
- Control group (No Intervention): Participants in this group will continue their usual activities.

INTERVENTIONS:
Other: Therapeutic dance — The protocol includes two sessions per week of therapeutic dance, during the months of October to May.
  Arms: Dance group

SUMMARY:
The goal of this clinical trial is to determine the effect of a therapeutic dance program developed in a school environment on different parameters of structure and function, activity and participation according to the ICF framework in children with functional diversity.

Researchers will compare the effects of eight months of therapeutic dance classes (consisting of two one-hour sessions per week) on ICF parameters to the effects of no intervention.

DETAILED DESCRIPTION:
This randomized clinical trial is designed to determine the effect of therapeutic dance developed in a school environment on different parameters of structure, function, activity, and participation according to the ICF framework in children with functional diversity. The study will include around 30 participants between the ages of 3 and 14.

Participants will be selected from five collaborating educational centers. Participants will be selected after an interview with teachers and after meeting the inclusion criteria. All families must sign an informed consent form allowing their child to participate. Each educational center will be randomly assigned to the intervention or control group.

The protocol includes two sessions per week from October to May. Each session lasts one hour. There will be two evaluations: one before the intervention begins and one at the end of the protocol. The primary outcomes include motor function, balance, walking speed, quality of life as perceived by patients and caregivers, and participation in daily activities.

This study adheres to the CONSORT guidelines and the Declaration of Helsinki, and it has been reviewed by an ethics committee.

ELIGIBILITY:
Inclusion Criteria:

* children with motor impairment
* aged between 3-14 years,
* who can cognitively follow simple tasks

Exclusion Criteria:

* having suffered a serious clinical condition or surgical intervention in the last 6 months.

Ages: 3 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
The Canadian Occupational Performance Measure (COPM). | Baseline (pre-intervention) and immediately post-intervention.
  Is an evidence-based outcome measure designed to capture a client's self-perception of performance in everyday living, over time.
Goal Attainment Scale (GAS). | Baseline (pre-intervention) and immediately post-intervention.
  Goal Attainment Scaling (GAS) is a method of scoring the extent to which patient's individual goals are achieved in the course of intervention.

SECONDARY OUTCOMES:
Quality of life with the Pediatric Quality of Life Inventory (PEDS QL) | Baseline (pre-intervention) and immediately post-intervention.
  A tool used to measure the health-related quality of life in children and adolescents, both with and without health conditions.
Gross Motor Function Measure (GMFM-88). | Baseline (pre-intervention) and immediately post-intervention.
  Is an assessment tool designed and evaluated to measure changes in gross motor function over time or with intervention in children with cerebral palsy.
Pediatric Balance Scale | Baseline (pre-intervention) and immediately post-intervention.
  The scale consists of 14 balance-related test items that are scored from 0 points (lowest function) to 4 points (highest function) with a maximum score of 56.
Timed up and go test (TUG) | Baseline (pre-intervention) and immediately post-intervention.
  This test involves a series of actions that assess an individual's mobility and balance. It requires the individual to rise from a seated position in a standard chair, walk a distance of three meters, turn around, walk back to the chair, and sit down again. The time it takes to complete this sequence is recorded.
Joint ranges | Baseline (pre-intervention) and immediately post-intervention.
  The joint ranges of the hip, knee and ankle in the three planes of movement will be carried out with a goniometer.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data may be shared with other researchers upon a reasonable request made to the project's principal investigator.
  Study Protocol will be published.
Supporting Information: Study Protocol, ICF